CLINICAL TRIAL: NCT02920840
Title: Brain-oscillation Synchronised Stimulation of the Prefrontal Cortex: Development and Validation of a Personalized Closed-loop TMS Protocol for the Treatment of Major Depression
Brief Title: Brain-oscillation Synchronised Stimulation of the Prefrontal Cortex
Acronym: BOSSFRONT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: BNP2016-03
Record Dates: First submitted 2016-09-26; First posted 2016-09-30 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2016-09

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Intermittent theta-burst stimulation (Active Comparator): Intervention: application of 200 TMS triplet bursts (at 100 Hz, inter-burst interval 200ms) over left dorsolateral prefrontal cortex
  Interventions: Device: Intermittent theta-burst stimulation
- Negative-peak-triggered-TMS (Experimental): Intervention: application of 200 brain-state dependent 100 Hz TMS triplet bursts triggered at the negative peak phase of the ongoing endogenous alpha-band oscillation (as detected by surface EEG over left dlPFC)
  Interventions: Device: Negative-peak-triggered-TMS
- Open-loop replay TMS (Active Comparator): Intervention: application of the same sequence of TMS pulses as in condition "Negative-peak-triggered-TMS", i.e. irrespective of ongoing brain state over left dlPFC
  Interventions: Device: Open-loop replay TMS

INTERVENTIONS:
Device: Intermittent theta-burst stimulation — see associated arm/group description
  Arms: Intermittent theta-burst stimulation
Device: Negative-peak-triggered-TMS — see associated arm/group description
  Arms: Negative-peak-triggered-TMS
Device: Open-loop replay TMS — see associated arm/group description
  Arms: Open-loop replay TMS

SUMMARY:
Combining TMS and EEG, this study investigates a personalized therapeutic non-invasive brain stimulation protocol in patients with major depression, whereby the timing of the TMS pulses is synchronized with the instantaneous phase of ongoing brain oscillations in order to modulate the inter-hemispheric left and right dorso-lateral prefrontal cortical brain network.

DETAILED DESCRIPTION:
Major depressive disorder is a severe psychiatric illness with a lifetime prevalence of about 8-16%. Many patients fail to achieve complete remission of symptoms under antidepressant medication, with about 10% of patients being chronically resistant to several psychopharmacological treatments. Development of alternative non-pharmacological treatments is therefore essential to improve patient care.

Repetitive transcranial magnetic stimulation (rTMS) offers therapeutic potential in this context. Current protocols apply high-frequency rTMS over left dorsolateral prefrontal cortex (DLPFC) to reverse the increased alpha-band oscillatory activity and cortical hypo-excitability in patients with depression. However, translation of rTMS therapy into routine clinical practice has been limited due to low efficacy and high inter-individual variability.

This study aims to optimize rTMS stimulation protocols for MDD by deterministically coupling the timing of TMS to the ongoing oscillatory neural activity in the underlying cortex as measured in real-time with high-density surface EEG. It is hypothesized that alpha phase-locked rTMS of the left DLPFC reverses increased alpha-band oscillatory activity and cortical hypo-excitability more efficiently than current open-loop rTMS protocols used in the treatment of MDD.

ELIGIBILITY:
Subject inclusion criteria

1. Subjects are between 18 to 65 years old
2. Subjects meet the Diagnostic and Statistical Manual of Mental Disorders (DSM)-4 criteria for current major depressive disorder (MDD), confirmed with the Structured Clinical Interview for DSM-4.
3. On the 21-item Hamilton Rating Scale for Depression (HRSD) subjects need to score 8 points or more.
4. Subject is in good physical and mental health. Subject understands the study procedures and agrees to participate in the study by giving written informed consent.
5. Subject is willing to comply with the study restrictions.

Subject exclusion criteria

1. Subject is under the age of legal consent.
2. Subject suffers of bipolar disorder.
3. Previous failure of nine or more electroconvulsive therapy treatments.
4. A current major depressive episode longer than 5 years.
5. A history of substance abuse or dependence within the past 2 years.
6. Subject suffers of antisocial or borderline personality disorder, active suicidal ideation with plan and/or intent.
7. Subject suffers of current symptoms of psychosis.
8. Subject has a history of seizure disorder.
9. Subject has a history of severe head injury with loss of consciousness.
10. Subject had a prior brain surgery, or any other major psychiatric or medical comorbidity.
11. Subjects with intake of pro-convulsive medication, e.g. imipramine, amitriptyline, doxepin, nortriptyline, maprotiline, chlorpromazine, clozapine, foscarnet, ganciclovir, ritonavir, amphetamines, cocaine, ecstasy, phencyclidine (PCP, angel's dust), ketamine, gamma-hydroxybutyrate (GHB), alcohol, theophylline, in accord with present consensus guidelines on safety, ethical considerations, and application of TMS in clinical practice and research (Rossi et al. 2009).
12. Subjects are allowed to continue their antidepressant medication, but must be on that medication for at least 2 months and on a stable dose for at least 4 weeks (6 weeks in the case of fluoxetine). Drug doses have to be kept constant during the study.
13. Patients with need of regular anxiolytic (e.g. benzodiazepine) treatment above 1 mg lorazepam/d.
14. Subjects are allowed to continue psychotherapy, but must be treated a minimum of 12 weeks prior to inclusion in the study, and type and frequency of psychotherapy must not be changed during the study period.
15. Subject has a cardiac pacemaker, implanted medication pump, intracardiac line, or acute, unstable cardiac disease.
16. Subject has an intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head (excluding the mouth) that cannot be safely removed.
17. Subject has participated in another study within 2 weeks prior to the first study visit.
18. Subject has contra-indications to MRI scans or does not agree that (1) the scans are obtained for research purposes only and will not be evaluated by a qualified neuroradiologist; if an abnormality is present, this may well not be noticed by the doctors, scientists and other staff involved in the study and handling the MRI data; and that (2) if any of the staff involved in the study do suspect a relevant abnormality to be present in any of the scans, they will reveal this to the subject so that a further diagnostic workup can be conducted outside of the study.
19. Subject is pregnant or trying to get pregnant.
20. Women of childbearing age should avoid.
21. Contraindications to an MRI

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-09; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in cortical excitability 30 minutes after the intervention | 30 minutes
  TMS-evoked EEG potentials from left dlPFC

SECONDARY OUTCOMES:
Change from baseline in EEG alpha power 30 minutes after the intervention | 30 minutes
  Left vs. right dlPFC relative spectral power in 8-12 Hz frequency band
Change from baseline in verbal working memory performance 30 minutes after the intervention | 30 minutes
  Verbal working memory task

OTHER OUTCOMES:
Change from baseline in mood on the Hamilton depression rating scale score 30 minutes after the intervention | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte Zrenner, MD, Study Director — University Neurology Hospital Tübingen; Florian Müller-Dahlhaus, MD, Study Director — University Neurology Hospital Tübingen; Ulf Ziemann, MD, Principal Investigator — University Neurology Hospital Tübingen; Andreas J Fallgatter, MD, Principal Investigator — University Psychiatry Hospital Tübingen; Surjo Soekadar, MD, Study Director — University Psychiatry Hospital Tübingen
Locations (1):
- University Neurology Hospital, Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided